CLINICAL TRIAL: NCT06715969
Title: Comparison of the Effects of Myofascial Release and Fascial Induction Therapy Techniques on Pain, Flexibility and Fascial Architecture.
Brief Title: Comparison of Two Different Fascial Treatments
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Doğan Burak Endamli (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Sponsor-Investigator, Doğan Burak Endamli, Expert physiotherapist, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HasanKalyon
Record Dates: First submitted 2024-11-19; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain, Mechanical
Keywords: low back pain; ultrasound; toracolumbal fascia
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Myofascial release will be applied to one group, miofascial induction treatment will be applied to the other group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- myofasyal indiction treatment (Active Comparator): MIT will be applied to the lumbal region by a physiotherapist trained and experienced in fascial treatments to patients in the MIT group. Applications 2 sessions per week, a total of 8 sessions will be applied, with an average of 20-25 minutes. The application principles of this technique will be as follows.
  * Induction of the lumbal interfacial triangle region (stroke application) (3 min)
  * Induction of the lumbal interfacial triangle region (deep induction application) (3 min)
  * Cross-hands myofascial induction (3 min)
  Interventions: Other: Myofascial Induction Techniques
- classıcal phsyotherapy (Active Comparator): 15 sessions of mictowave diathermy (MDD), Vacuum Interference, Infraruj and Classic waist exercise program will be applied to patients in this group.
  Interventions: Other: classıcal phsyotherapy
- Myofacial ReleaseTechniques (Active Comparator): Separate techniques will be applied to the parts of the thoracolumbal fascia that surround the erector spina, quadratus lumborum, latissimus dorsi muscles and extend in that direction to patients in the MFR group. Techniques will continue for 180 seconds, tissue shift will be carried further as relaxation is achieved. Applications Total 8 sessions will be applied twice a week by an experienced physiotherapist.
  Interventions: Other: Myofascial Release Techniques

INTERVENTIONS:
Other: Myofascial Release Techniques — Separate techniques will be applied to the parts of the thoracolumbal fascia that surround the erector spina, quadratus lumborum, latissimus dorsi muscles and extend in that direction to patients in the MFR group. Techniques will continue for 180 seconds, tissue shift will be carried further as relaxation is achieved. Applications Total 8 sessions will be applied twice a week by an experienced physiotherapist.
  Arms: Myofacial ReleaseTechniques
Other: Myofascial Induction Techniques — MIT will be applied to the lumbal region by a physiotherapist trained and experienced in fascial treatments to patients in the MIT group. Applications 2 sessions per week, a total of 8 sessions will be applied, with an average of 20-25 minutes. The application principles of this technique will be as follows.
  * Induction of the lumbal interfacial triangle region (stroke application) (3 min)
  * Induction of the lumbal interfacial triangle region (deep induction application) (3 min)
  * Cross-hands myofascial induction (3 min)
  Arms: myofasyal indiction treatment
Other: classıcal phsyotherapy — 15 sessions of mictowave diathermy (MDD), Vacuum Interference, Infraruj and Classic waist exercise program will be applied to patients in this group.
  Arms: classıcal phsyotherapy

SUMMARY:
The aim of this study is to compare the different effects of two different fascial treatments on pain, flexibility and Asian architecture.

2 different groups 8 sessions, two different fascial treatments will be applied in accordance with the intake criteria, the individuals will be re-evaluated before the treatment, after 8 sessions of treatment and 3 months after the end of the study.

DETAILED DESCRIPTION:
Chronic low back pain is a disease that causes the loss of working days in the world, causes significant disability and health costs, and cannot be fully diagnosed. It ranks second among the job loss factors and is considered the most important factor affecting the decline in production.

Until recent years, conservative treatment of all types of low back pain included bed rest for a certain period of time. This situation has changed over time with studies, and today's treatment is to gradually increase the level of activity according to the person's level with minimal bed rest.

Chronic low back pain is seen as a disorder that 70% of people can experience at least once in their lives. Today, it is one of the most common and expensive syndromes of modern times, reaching a rate of 80% in Europe. The participants experiencing the negative effects of chronic low back pain has disadvantages such as health and medical research expenses for the community, while experiencing pain, decreased daily living activities, decreased work productivity or disappearance.

There are no regional, national and international guidelines for the treatment of chronic low back pain. There is no strong recommendation for a specific physiotherapy approach yet. Studies to understand the pathophysiological mechanisms that lead to this focus on the structural pathology of the spine and related tissues, neuropsychosocial factors and motor control abnormalities. On the other hand, the fascia of the lumbal region received little attention.

Several researchers have suggested that fascias may play a role in the pathophysiology of LBP. In one study, it was seen that the thoracolumbal fascia (TLF) was thicker in the ultrasound image of people who experienced LBP than in normal people. Recent studies have shown a relationship between LBP and facial tissue. However, there is no treatment program for this.

Each body structure is surrounded by fascia, and for every tissue and organ, fascias form and create a continuity that provides function. Each region of the human body should be accepted as a functional unit in communication with each other with the fascial continuity. Facial tissue is evenly distributed and interacts with nerves and veins in particular. It forms layers in the depths of internal organs, bones and muscles and forms a three-dimensional mechanical and metabolic matrix. Therefore, the fascia becomes an organ that can affect a person's health. The continuity of the fascia in the body and the mechanical role of fibroblasts, the ability to communicate with each other, strengthens the belief that the fascia has a similar integration in the nervous system.

The Myofascial Release Technique (MFR) is one of the manual techniques used to increase the lengthenability of soft tissues or to restore normal length in limited fascia or muscles by providing a continuous stretch or compression to target tissues. MFR method is a method applied under the skin without slipping on the skin. The face matrix responds to 4 mechanoreceptors (golgi, paccini, ruffini and intersitial). The MFR stimulates these mechanoreceptors by increasing the awareness of touch and kinesthetics, applying pressure-sensitive techniques, and then applying constant pressure to release the restricted fascia. As the tissue relaxes, it stretches and the patient begins to loosen on its own, other mechanical receptors are stimulated by this movement. The MFR also allows collagen and elastin fibers to be rearranged to a more suitable resting length by applying biomechanical energy or by pressure from energy.

Myofacial Induction Technique (MIT) is a method used in physiotherapy that focuses on the restoration of modified phased tissues. In a healthy body, the facial system provides flexibility and coordination of movements. With MIT, the healing of a region is achieved by changing the tissue dynamics due to the mechanical tension of the region. Fascia acts as a space-sensitive system. During treatment, the clinic stretches or compresses a specific body area to transmit a low-intensity mechanical stimulation. This input creates changes that spread to body systems at the molecular level. Chemically, metabolic and physiologically, it creates mutual reactions in the body. MIT is a therapy concept that focuses on optimizing function and balance within the facial system. The approach aims at local healing, improving global dynamics and painless body use. The treatment protocol is divided into 2 stages, superficial techniques and deep procedures. Surface procedures are intended for surface and/or local restrictions that can be directly detected by palpation. Deep myofascial induction treatment, on the other hand, is a method that eliminates the limitations of the movements applied to the myofascial system and the pressures used in three dimensions.

When the literature was examined, fascia treatments in people with chronic low back pain were investigated, it was found to be effective, but it was found that more than one technique was not compared. In addition, the instantaneous or short-term effects of fascia treatments have always been taken into account. In addition, the information that the tocolumbal fascia surrounds many muscles and also covers them has been neglected. These limitations have led us to do this job. In the light of this information, the aim of our study is to determine the most effective fascia treatment and to present the literature as a result of the treatments of people with chronic low back pain in Gaziantep.

Our study will be planned as a randomized controlled study. Our most legal goal is that our treatment method applied manually in our study is morphological changes in the body by looking at it with ultrasound. It is predicted that our study will shed light on the studies to be carried out on fascial therapies, which have come to the fore in the last few years and whose importance is increasing every year.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 35-60 years old
* Patients with low back pain for at least 3 months
* Patients with pain 4 and above according to VAS
* Having not received FTR and manual therapy for the last 3 months
* Those who have not received medical treatment for the last 3 months and those who will not

Exclusion Criteria:

* Those with a history of back and spine surgery
* Patients with a history of trauma
* Those with instable neurological findings
* Having a pathology such as hernia and root pressure in the lumbal region
* Regular users of analgesic and anti-inflammatory drugs
* Communication problem that will prevent the implementation of evaluations and/or treatment program

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
pain | From enrollment to the end of treatment at 4 weeks
  We expect a decrease in pain at the end of 4 weeks. We expect a decrease in the value of the visual analog scale (VAS). According to this scale, it shows 10 very severe pains and 0 pains. We look at the VAS values of people both before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: kezban bayramlar, profesör, Study Director — Hasan Kalyoncu University
Locations (1):
- MMT Amerikan tıp merkezi, Gaziantep, sehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chamorro Comesana A, Suarez Vicente MD, Docampo Ferreira T, Perez-La Fuente Varela MD, Porto Quintans MM, Pilat A. Effect of myofascial induction therapy on post-c-section scars, more than one and a half years old. Pilot study. J Bodyw Mov Ther. 2017 Jan;21(1):197-204. doi: 10.1016/j.jbmt.2016.07.003. Epub 2016 Jul 18. PMID 28167179